CLINICAL TRIAL: NCT06211309
Title: Evaluation of Anti-plaque and Anti-inflammatory Effects of Green Tea and Salvadora Persica L. in Patients With Gingivitis
Brief Title: The Effects of Green Tea and Salvadora Persica L. in Patients With Gingivitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Aliaa Saeed Salman, principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 857623
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gingivitis
Keywords: Dental plaque; Salvadora; Green tea; Mouthwash; Clinical trial
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- co.mouthwash (Active Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Drug: co.mouthwas
- Kin mouthwash (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Kin
- Distilled water (Placebo Comparator): 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: co.mouthwas — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Other Names: co
  Arms: co.mouthwash
Other: Kin — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Kin mouthwash
Other: Distilled water — 15ml twice a day, rinse for 30sec refrain from eating or drinking for 30min
  Arms: Distilled water

SUMMARY:
Gingivitis is an inflammatory condition of the gingival tissue, most commonly caused by bacterial infection.The plaque control is considered the most important preventive factor concerning caries, gingivitis, and periodontitis Mechanical means of plaque control, e.g. tooth brushing, flossing and use of other mechanical devices are the most commonly used methods. However, ideal plaque control solely by mechanical means requires a significant effort and is difficult to achieve.This has led to the introduction of chemical methods of plaque control using antimicrobial agentsMore specifically, chemotherapeutic agents with antimicrobial properties, such as 0.12% chlorhexidine (CHX).chx has side effects encourage the need to develop alternative mouthwashes with similar efficacy but without these issues.hence the mouthwash enriched with a combination of aqueous extracts of Salvadora persica L. and green tea used as a substitution to CHX with minimal side effects .The objective of this study was to investigate the efficacy of the combination of Gt aqueous extract and Sp aqueous extract in reducing plaque buildup and gingivitis for 4 weeks duration.

DETAILED DESCRIPTION:
Gingivitis is an inflammatory condition of the gingival tissue, most commonly caused by bacterial infection. Unlike periodontitis, there is no attachment loss and therefore no migration of the junctional epithelium. The condition is restricted to the soft-tissue area of the gingival epithelium and connective tissue.Gingivitis is caused by the microbial plaque deposits located in or close to the gingival sulcus).

The plaque control is considered the most important preventive factor concerning caries, gingivitis, and periodontitis Mechanical means of plaque control, e.g. tooth brushing, flossing and use of other mechanical devices are the most commonly used methods. However, ideal plaque control solely by mechanical means requires a significant effort and is difficult to achieve.This has led to the introduction of chemical methods of plaque control using antimicrobial agentsMore specifically, chemotherapeutic agents with antimicrobial properties, such as 0.12% chlorhexidine (CHX), have been proposed as an adjunct to the standard oral hygiene protocol. chx has side effects encourage the need to develop alternative mouthwashes with similar efficacy but without these issues.

Hence the mouthwash enriched with a combination of aqueous extracts of Salvadora persica L. and green tea used as a substitution to CHX with minimal side effects .

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged more than 15 years-old who will volunteer to participate.
2. Participants who were apparently systemically healthy.
3. Not taking antibiotic and anti-inflammatory drugs in the last three months
4. Patients having generalized gingivitis with intact periodontium in which they have more than 30% bleeding sites with no PPD >3 mm with no clinical attachment loss according to criteria proposed by

Exclusion Criteria:

1. Those with history of systemic chronic disease, immunocompromised patients.
2. Those currently using any mouthwash.
3. Those on antibiotic therapy, anti-inflammatory medications or NSAID during the study and at the last 3 months before the study.
4. Those having a history of hypersensitivity to any product used in the present study.
5. Those having periodontitis.
6. Those who smoker or alcoholism.
7. handicapped patient or patients with limited manual dexterities.
8. pregnant , lactating women or taking contraceptive pills.
9. Subjects wearing orthodontic appliances or removable dentures.
10. patients unwilling to participate in study.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
change in plaque index | 0-30 days
  Mean amount plaque between different comparators. Mean amount plaque between different comparators as anti-plaque agent after rinsing with different comparators using means of modified quigely hein plaque index[ Turesky ,1970

SECONDARY OUTCOMES:
Change in BOP score | 0-30 Days
  For recording BOP score, the periodontal probe was inserted with gentle force into the sulcus/pocket until minimal resistance was felt. The probing force presumably was ranging between 20 to 25g. The examination started from the distal surface of the right upper 7 moving mesially to measure all the existing teeth. For each tooth, 6 surfaces were examined; the surface that displayed bleeding on probing was scored 1 and the surface with no bleeding was scored 0
change in Gingival index | 0-30 days
  Subjects will undergo the measurement of gingival index according to Loe & Silness, designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency and bleeding on probing. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva. Data will be collected based on four possible clinical conditions: 0=Normal gingiva1=Mild Inflammation-Slight change in color, Slight odema. No bleeding on probing2=Moderate inflammation-redness,odema and glazing. Bleeding on probing 3=Sever inflammation-marked redness and edema.Ulceration.Tendency to spontaneous bleeding.
Mean relative change in cytokine interleukin-6 level in salivary Fluid | 0-30 days
  Mean relative change in cytokine interleukin-6 level in salivary Fluid after washing with different mouthwash from baseline at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aliaa, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided